CLINICAL TRIAL: NCT01798680
Title: Trial of Vitamin D in HIV Progression
Acronym: TOV4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Management and Development for Health (MDH) (Unknown)
Responsible Party: Principal Investigator, Wafaie Fawzi, Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01DK098075 (NIH)
Record Dates: First submitted 2013-02-21; First posted 2013-02-26 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (cholecalciferol) (Experimental)
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — Supplements containing 50,000 IU of vitamin D3 (cholecalciferol) taken orally once per week for 4 weeks (weeks 0, 1, 2, 3) followed by 2,000 IU of vitamin D3 (cholecalciferol) supplements taken orally once per day starting at 4 weeks until study discharge at 12 months
  Arms: Vitamin D3 (cholecalciferol)
Other: Placebo — Placebo pills taken once weekly for 4 weeks (weeks 0, 1, 2, 3) followed by placebo pills taken orally once per day starting at 4 weeks until study discharge at 12 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of vitamin D3 (cholecalciferol) supplementation on HIV progression and incidence of pulmonary tuberculosis among HIV-positive Tanzanian adult men and women initiating highly active antiretroviral therapy (HAART).

DETAILED DESCRIPTION:
HIV-infected adults initiating antiretroviral therapy in resource-limited settings experience high mortality, pulmonary tuberculosis, and other comorbidity rates during the first year of HIV treatment. Observational studies have shown low vitamin D is a risk factor for HIV progression and incidence of pulmonary tuberculosis among adults initiating HAART; however, whether this relationship is causal and if vitamin D supplementation starting at HAART initiation can improve health outcomes has not been determined. This study is a randomized, double-blind, placebo-controlled trial conducted to examine the effect of vitamin D3 supplementation on morality and pulmonary tuberculosis for adults initiating HAART. Participants are HIV-positive Tanzanian men and women aged 18 years and older, who are initiating HAART at the time of randomization whose baseline 25-hydroxyvitamin D (25(OH)D) concentration is <30ng/mL. Eligible individuals are randomized to receive a) a vitamin D3 regimen consisting 50,000 IU of vitamin D3 taken orally once per week for 4 weeks (weeks 0, 1, 2, 3) followed by 2,000 IU of vitamin D3 supplements taken orally once per day starting at 4 weeks until study discharge at 12 months or b) placebo pills taken once weekly for 4 weeks (weeks 0, 1, 2, 3) followed by placebo pills taken daily starting at 4 weeks until study discharge. Participants will be followed for 12 months after ART initiation.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Men or Women
* 18 Years of Age or older
* Initiating HAART at time of randomization
* 25(OH)D concentration <30 ng/mL at HAART initiation

Exclusion Criteria:

* Pregnant Women
* Enrolled in another micronutrient trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
All-cause death | within 12 months after randomization
Pulmonary tuberculosis | within 12 months after randomization

SECONDARY OUTCOMES:
CD4+ T-cell count | 6 and 12 months after randomization
Physician diagnosis of comorbidities | within 12 months after randomization
Parathyroid hormone (PTH) | 1, 6, and 12 months after randomization
Alkaline phosphatase (ALP) | 1, 6, and 12 months after randomization
>10% weight loss | monthly from month 1 to month 12
Wasting (BMI <18.5 kg/m2) | monthly from month 1 to month 12
Hypercalcemia | 1, 6, and 12 months after randomization
Physical activity | 6 and 12 months after randomization
Immunologic biomarker levels (IL-2, IL-12, IFN-γ, and cathelicidin) | 1, 6, and 12 months after randomization
Depression and anxiety scores | 6 and 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MBBS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH); Ferdinand M Mugusi, MD, Principal Investigator — Management and Development for Health (MDH)
Locations (1):
- Management and Development for Health (MDH), Dar es Salaam, Tanzania

REFERENCES:
- [Background] Sudfeld CR, Mugusi F, Aboud S, Nagu TJ, Wang M, Fawzi WW. Efficacy of vitamin D3 supplementation in reducing incidence of pulmonary tuberculosis and mortality among HIV-infected Tanzanian adults initiating antiretroviral therapy: study protocol for a randomized controlled trial. Trials. 2017 Feb 10;18(1):66. doi: 10.1186/s13063-017-1819-5. PMID 28183335
- [Derived] Muhihi A, Fawzi WW, Aboud S, Nagu TJ, Ulenga N, Wang M, Mugusi F, Sudfeld CR. Cholecalciferol Supplementation Does Not Affect the Risk of HIV Progression, Viral Suppression, Comorbidities, Weight Loss, and Depression among Tanzanian Adults Initiating Antiretroviral Therapy: Secondary Outcomes of a Randomized Trial. J Nutr. 2022 Aug 9;152(8):1983-1990. doi: 10.1093/jn/nxac096. PMID 35460249
- [Derived] Sudfeld CR, Mugusi F, Muhihi A, Aboud S, Nagu TJ, Ulenga N, Hong B, Wang M, Fawzi WW. Efficacy of vitamin D3 supplementation for the prevention of pulmonary tuberculosis and mortality in HIV: a randomised, double-blind, placebo-controlled trial. Lancet HIV. 2020 Jul;7(7):e463-e471. doi: 10.1016/S2352-3018(20)30108-9. PMID 32621874